CLINICAL TRIAL: NCT00955487
Title: Examining the Use of Non-Invasive Inhaled Nitric Oxide to Reduce Chronic Lung Disease in Premature Newborns
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06-0124; 5P50HL084923 (NIH); 5 P50 HL084923-030001
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Premature Newborns; Inhaled Nitric Oxide
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Nitrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Nitric Oxide (iNO) (Experimental): Participants will receive a low concentration of iNO until they are 30 weeks corrected gestational age or for 14 days if they were born at 29 weeks or more.
  Interventions: Drug: Inhaled Nitric Oxide (iNO)
- Nitrogen (placebo) (Placebo Comparator): Participants will receive nitrogen (placebo) while in the hospital.
  Interventions: Drug: Nitrogen (placebo)

INTERVENTIONS:
Drug: Inhaled Nitric Oxide (iNO) — iNO will be delivered using the iNOVent device to provide 10 ppm proximally (yielding approximately 5 ppm to the posterior pharynx).
  Arms: Inhaled Nitric Oxide (iNO)
Drug: Nitrogen (placebo) — Nitrogen will be delivered using the iNOVent device to provide 10 ppm proximally (yielding approximately 5 ppm to the posterior pharynx).
  Arms: Nitrogen (placebo)

SUMMARY:
Bronchopulmonary dysplasia (BPD) is a serious lung condition that affects premature newborns. The condition involves abnormal development of lung tissue and is characterized by inflammation and scarring in the lungs. Treatment with inhaled nitric oxide (iNO) may reduce the incidence of BPD and another commonly associated condition called pulmonary hypertension, which is high blood pressure in the vessels carrying blood to the lungs.. This study will determine if early treatment with low-dose iNO reduces the incidence of BPD, pulmonary hypertension, and death in premature newborns.

DETAILED DESCRIPTION:
BPD is a serious lung condition that primarily affects premature newborns and newborns with low birth weights. iNO has been proven to be a safe and effective treatment for pulmonary hypertension and hypoxemic respiratory failure-both of which are abnormal lung conditions-in full-term newborns. However, in babies born prematurely, the effects of iNO on lung function are not well defined. Also, previous studies have mainly examined whether iNO reduces the incidence of BPD in newborns who are on mechanical ventilation. However, intubation and mechanical ventilation of premature newborns is now increasingly being avoided, and non-invasive support, including the use of nasal continuous positive airway pressure (NCPAP), is being used. Early treatment with low-dose iNO may reduce the incidence of BPD in premature newborns who do not require mechanical ventilation and intubation after delivery. The purpose of this study is to determine if low-dose, non-invasive iNO reduces the risk of BPD, pulmonary hypertension, and death in premature newborns who do not require mechanical ventilation.

This study will enroll premature newborns who require extra oxygen but do not require intubation or mechanical ventilation for respiratory failure in the first 72 hours of life. Participants will be randomly assigned to receive low-dose, non-invasive iNO or nitrogen (placebo) during their hospital stay. While hospitalized, participants' heart rate, blood oxygen level breathing rate, blood pressure, and medications will be monitored, and blood collection will occur at various times. Monitoring will continue until participants are 30 weeks corrected gestational age or for at least 14 days if participants are born at 29 weeks or more. All participants will undergo an ultrasound of the head when they are 7 days, 28 days, and 36 weeks of age. They will undergo an echocardiogram, which is an ultrasound of the heart, at 7 and 21 days of age and 4 weeks before the original expected due date. A chest x-ray will be performed before hospital discharge, and a breathing status test will be performed either 4 weeks before participants' original expected due date or before hospital discharge. Follow-up study visits will occur at Years 1 and 2, and will include a physical examination and developmental and behavioral testing. Another echocardiogram will also be performed at the Year 1 visit.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight of 500-1250 grams and gestational age of less than 34 weeks
* Age at enrollment is less than 72 hours
* Supplemental oxygen or 21% requirement by nasal cannula or NCPAP only

Exclusion Criteria:

* Presence of structural heart disease (other than patent ductus arteriosus, atrial septal defect less than 1 cm, or muscular ventricular septal defect less than 2 mm)
* Presence of lethal congenital anomaly
* Participating in another concurrent experimental study
* Requires mechanical ventilation in the first 72 hours of life (patients are not excluded if they are intubated briefly but they must be extubated at the time of consent and study entry prior to 72 hours of life)

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2007-01; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kinsella, MD, Principal Investigator — Chidlren's Hospital and University of Colorado Hospital
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, San Diego, California
  - Children's Hospital and University Colorado Hospital, Aurora, Colorado
  - Anne and Robert H. Lurie Children's Hospital of Chicago and Northwestern Memorial Hospital, Chicago, Illinois
  - Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt Children's Hospital, Nashville, Tennessee

REFERENCES:
- [Derived] Kinsella JP, Cutter GR, Steinhorn RH, Nelin LD, Walsh WF, Finer NN, Abman SH. Noninvasive inhaled nitric oxide does not prevent bronchopulmonary dysplasia in premature newborns. J Pediatr. 2014 Dec;165(6):1104-1108.e1. doi: 10.1016/j.jpeds.2014.06.018. Epub 2014 Jul 22. PMID 25063725

RESULTS

PARTICIPANT FLOW:
Groups:
- 500-749g Inhaled Nitric Oxide (iNO): Participants weighing between 500 and 749 grams received a low concentration of iNO until they were 30 weeks corrected gestational age or for 14 days if they were born at 29 weeks or more.
  iNO was initiated at 10ppm to yield a minimum of 5ppm to the posterior pharynx.
- 500-749g Placebo (Nitrogen): Participants weighing between 500 and 749 grams received Placebo (Nitrogen) until they were 30 weeks corrected gestational age or for 14 days if they were born at 29 weeks or more.
  Placebo was initiated at 10ppm to yield a minimum of 5ppm to the posterior pharynx.
- 750-999g Inhaled Nitric Oxide (iNO): Participants weighing between 750-999 grams received a low concentration of iNO until they were 30 weeks corrected gestational age or for 14 days if they were born at 29 weeks or more.
  iNO was initiated at 10ppm to yield a minimum of 5ppm to the posterior pharynx.
- 750-999g Placebo (Nitrogen): Participants weighing between 750 and 999 grams received Placebo (Nitrogen) until they were 30 weeks corrected gestational age or for 14 days if they were born at 29 weeks or more.
  Placebo was initiated at 10ppm to yield a minimum of 5ppm to the posterior pharynx.
- 1000-1250g Inhaled Nitric Oxide (iNO): Participants weighing between 1000 and 1250 grams received a low concentration of iNO until they were 30 weeks corrected gestational age or for 14 days if they were born at 29 weeks or more.
  iNO was initiated at 10ppm to yield a minimum of 5ppm to the posterior pharynx.
- 1000-1250g Placebo (Nitrogen): Participants weighing between 1000 and 1250 grams received Placebo (Nitrogen) until they were 30 weeks corrected gestational age or for 14 days if they were born at 29 weeks or more.
  Placebo was initiated at 10ppm to yield a minimum of 5ppm to the posterior pharynx.
Period: Overall Study
Arm/Group | 500-749g Inhaled Nitric Oxide (iNO) | 500-749g Placebo (Nitrogen) | 750-999g Inhaled Nitric Oxide (iNO) | 750-999g Placebo (Nitrogen) | 1000-1250g Inhaled Nitric Oxide (iNO) | 1000-1250g Placebo (Nitrogen)
Started | 10 | 9 | 17 | 21 | 32 | 35
Completed | 10 | 9 | 17 | 21 | 32 | 35
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inhaled Nitric Oxide (iNO): Participants will receive a low concentration of iNO until they are 30 weeks corrected gestational age or for 14 days if they were born at 29 weeks or more.
  Inhaled Nitric Oxide (iNO) will be delivered using the iNOVent device to provide 10 ppm proximally (yielding approximately 5 ppm to the posterior pharynx).
- Placebo (Nitrogen): Participants will receive Placebo until they are 30 weeks corrected gestational age or for 14 days if they were born at 29 weeks or more.
  Placebo will be delivered using the iNOVent device to provide 10 ppm proximally (yielding approximately 5 ppm to the posterior pharynx).
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen) | Total
Number analyzed (Participants) | 59 | 65 | 124
Age, Customized [Mean (Standard Deviation); unit: Weeks]
  Gestational Age at Baseline | 27.5 (1.6) | 27.3 (1.8) | 27.4 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 24 | 31 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Mother's race/ethnic group
  Participants
    White | 48 | 48 | 96
    Black | 8 | 11 | 19
    Other | 3 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 65 | 124

OUTCOME MEASURES:

1. Primary Outcome: Combined Endpoint of Bronchopulmonary Dysplasia (BPD) or Mortality
Description: Number of participants that developed bronchopulmonary dysplasia and/or that died
Time Frame: Week 36 or earlier, if participants are discharged from the hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 65
Participants
  Death | 1 | 2
  Bronchopulmonary Dysplasia (BPD) | 24 | 25
  Death/BPD | 25 | 26
  No Death or BPD | 9 | 12

2. Primary Outcome: Combined Endpoint of Bronchopulmonary Dysplasia (BPD) or Mortality Stratified by Birth Weight
Description: Number of participants that developed bronchopulmonary dysplasia and/or that died, stratified by birth weight (grams)
Time Frame: Randomization to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | 500-749g Inhaled Nitric Oxide (iNO) | 500-749g Placebo (Nitrogen) | 750-999g Inhaled Nitric Oxide (iNO) | 750-999g Placebo (Nitrogen) | 1000-1250g Inhaled Nitric Oxide (iNO) | 1000-1250g Placebo (Nitrogen)
Number analyzed (Participants) | 10 | 9 | 17 | 21 | 32 | 35
Participants
  Death | 0 | 2 | 1 | 0 | 0 | 0
  BPD | 3 | 4 | 8 | 6 | 13 | 15
  Death/BPD | 3 | 5 | 9 | 6 | 13 | 15

3. Secondary Outcome: Severity of Bronchopulmonary Dysplasia (BPD)
Description: Assessment of the severity of BPD as defined by the oxygen reduction test
Time Frame: 36 weeks corrected gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 62
Participants
  None | 35 | 37
  Mild | 2 | 9
  Moderate | 20 | 12
  Severe | 2 | 4

4. Secondary Outcome: Need for Mechanical Ventilation
Description: Number of participants who required endotracheal intubation and mechanical ventilation
Time Frame: Anytime after randomization up to 36 weeks corrected gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 65
Participants
  Required Mechanical Ventilation | 13 | 15
  Did not require mechanical ventilation | 46 | 50

5. Secondary Outcome: Total Ventilation Days
Description: Of those participants who required mechanical ventilation, the total number of days receiving ventilation
Time Frame: After randomization up until hospital discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 65
Days | 9.7 (29) | 8.4 (12)

6. Secondary Outcome: Necrotizing Enterocolitis (NEC)
Description: Number of participants diagnosed with necrotizing enterocolitis
Time Frame: After randomization through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 65
Participants | 5 | 10

7. Secondary Outcome: Symptomatic PDA Requiring Medical Treatment
Description: Number of participants with a symptomatic PDA that required medical treatment
Time Frame: From randomization until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 65
Participants | 1 | 2

8. Secondary Outcome: Symptomatic PDA Requiring Surgical Ligation
Description: Number of participants with symptomatic PDA that required surgical ligation
Time Frame: Randomization through discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 65
Participants | 3 | 8

9. Secondary Outcome: Threshold Retinopathy of Prematurity (ROP)
Description: Threshold ROP defined as requiring interventional therapy
Time Frame: Randomization to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 65
Participants | 3 | 4

10. Secondary Outcome: Severe Intracranial Hemorrhage
Description: Number of participants that developed severe intracranial hemorrhage (grade 3-4)
Time Frame: Randomization to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 65
Participants | 2 | 4

11. Secondary Outcome: Sepsis
Description: Number of participants that developed sepsis
Time Frame: Randomization to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 65
Participants | 13 | 14

12. Other Pre Specified Outcome: Days in Hospital
Description: Length of stay of participants
Time Frame: From birth to hospital discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
Number analyzed (Participants) | 59 | 65
Days | 75 (32) | 75 (29)

ADVERSE EVENTS:
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo (Nitrogen)
All-Cause Mortality (participants affected / at risk) | 2/59 | 4/65
Serious Adverse Events (participants affected / at risk) | 27/59 | 42/65
Other Adverse Events (participants affected / at risk) | 0/59 | 0/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (iNO) (N=59) | Placebo (Nitrogen) (N=65)
Necrotizing enterocolitis (Gastrointestinal disorders) | 5 (5) | 10 (10)
Symptomatic PDA (Cardiac disorders) | 1 (1) | 2 (2) — Medical treatment
Symptomatic PDA (Cardiac disorders) | 3 (3) | 8 (8) — surgical treatment
Threshold ROP (Eye disorders) | 3 (3) | 4 (4)
Severe ICH (Nervous system disorders) | 2 (2) | 4 (4)
Sepsis (Infections and infestations) | 13 (13) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No